CLINICAL TRIAL: NCT05424926
Title: Switch From Intravenous to Subcutaneous Infliximab (REMSIMA®) in Clinical Practice in the Rheumatology Department of Cochin Hospital
Brief Title: Sub-cutaneous Infliximab in Inflammatory Rheumatic Disease
Acronym: SIC2
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211217; 2021-A02060-41 (Other: ANSM)
Record Dates: First submitted 2021-12-06; First posted 2022-06-21 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis; Spondyloarthritis; Psoriatic Arthritis
Keywords: Chronic inflammatory diseases; Biosimilar; Sub-cutaneous route
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Arthritis, Psoriatic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients
  Interventions: Other: collection of clinical parameters and blood sample

INTERVENTIONS:
Other: collection of clinical parameters and blood sample — * A baseline visit, with collection of clinical parameters and blood sample to measure anti-infliximab antibodies and infliximab trough levels.
  * Follow-up visits at 3 months (in outpatient clinic for clinical evaluation), 6 months and 12 months (in day hospitalization for clinical evaluation and blood sample collection for ADA detection and infliximab trough level measurement).

SUMMARY:
TNFα inhibitors have revolutionized the management of patients suffering from inflammatory diseases in the field of rheumatology. Infliximab remains widely used in France, and infliximab biosimilars have been routinely used since 2015 in Cochin Hospital with an interchangeability strategy validated by two real life studies. REMSIMA® 120 mg is the first authorized subcutaneous (SC) form of infliximab to be administered at a fixed dose of 120 mg every 2 weeks. Scarce information is available regarding the safety and efficacy of proposing a switch from IV infliximab to SC REMSIMA® in the subsets of patients suffering from different rheumatic diseases in daily care. The primary objective of the SIC2 study will be determine the retention rate of Remsima SC at 6 months. The investigators will recruit adult patients with rheumatoid arthritis, spondyloarthritis, psoriatic arthritis.

DETAILED DESCRIPTION:
TNFα inhibitors have revolutionized the management of patients suffering from inflammatory diseases in the field of rheumatology. Infliximab remains widely used in France, and infliximab biosimilars have been routinely used since 2015 in Cochin Hospital with an interchangeability strategy validated by two real life studies. REMSIMA® 120 mg is the first authorized subcutaneous (SC) form of infliximab to be administered at a fixed dose of 120 mg every 2 weeks. Scarce information is available regarding the safety and efficacy of proposing a switch from IV infliximab to SC REMSIMA® in the subsets of patients suffering from different rheumatic diseases in daily care. The primary objective of the SIC2 study will be determine the retention rate of Remsima SC at 6 months. The investigators will recruit adult patients with rheumatoid arthritis, spondyloarthritis, psoriatic arthritis. Main inclusion criteria will be patients who have received at least 3 IV infliximab infusions and suffer from chronic inflammatory rheumatic condition with the absence of disease flare / progressive disease preventing the continuation of infliximab. The primary endpoint will be the percentage of patients who have agreed to receive SC REMSIMA® and who continued this treatment for at least 3 months. Secondary objectives will be the reasons of switching or not to Remsima, the need for patients to be re-established on iv infliximab, SC Remsima® discontinuation and adherence, changes in disease activity between the inclusion visit and the last visit, the safety profile of sc remsima®, the immunogenicity profile of sc remsima®.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older
* Patients who has received at least 3 IV infliximab infusions and suffer from chronic inflammatory rheumatic condition
* Absence of disease flare / progressive disease preventing the continuation of infliximab
* Patient affiliated to national insurance

Exclusion Criteria:

* Any patient whose doctor considers that he will not be able to comply with the obligations of the trial
* Patients under curatorship or tutorship
* Pregnant women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who have agreed to receive SubCutaneous (SC) REMSIMA® and who continued this treatment for at least 6 months. | Month 6
  Therapeutic maintenance of SC REMSIMA® at 6 months, defined by the percentage of patients who have agreed to receive SC REMSIMA® and who continued this treatment for at least 6 months.

SECONDARY OUTCOMES:
Percentage of patients switching or not switching to remsima® SC | Day 0
  Percentage of patients switching or not switching to remsima® sc (refusal, need to maintain iv, etc.) with the analysis of the reasons of non-switching
Number of patients who requested to be re-established on intravenous(IV) infliximab | Month 3
  Number of patients who requested to be re-established on iv infliximab
Number of patients who requested to be re-established on iv infliximab | Month 6
  Number of patients who requested to be re-established on iv infliximab
Number of patients who requested to be re-established on iv infliximab | Month 12
  Number of patients who requested to be re-established on iv infliximab
Number of sc remsima® discontinuation | Month 3
  Number of sc remsima® discontinuation
Questionnaire about reasons explaining Remsina discontinuation | Month 3
  Reasons of sc remsima® discontinuation
Number of sc remsima® discontinuation | Month 6
  Number of sc remsima® discontinuation
Questionnaire about reasons explaining Remsina discontinuation | Month 6
  Reasons of sc remsima® discontinuation
Number of sc remsima® discontinuation | Month 12
  Number of sc remsima® discontinuation
Questionnaire about reasons explaining Remsina discontinuation | Month 12
  Reasons of sc remsima® discontinuation
Number of missing SC injections | Month 3
  Number of missing SC injections
Questionnaire about reasons explaining the missing of a scheduled Remsina injection | Month 3
  Reasons of missing SC injections
Number of missing SC injections | Month 6
  Number of missing SC injections
Questionnaire about reasons explaining the missing of a scheduled Remsina injection | Month 6
  Reasons of missing SC injections
Number of missing SC injections | Month 12
  Number of missing SC injections
Questionnaire about reasons explaining the missing of a scheduled Remsina injection | Month 12
  Reasons of missing SC injections
Frequencies of serious adverse effects | Month 3
  Safety profile of sc remsima®
Frequencies of serious adverse effects | Month 6
  Safety profile of sc remsima®
Frequencies of serious adverse effects | Month 12
  Safety profile of sc remsima®
Percentage of positive ADA | Month 6
  Immunogenicity profile of sc remsima®, consisting on the percentage of positive ADA at 6 months
Percentage of positive ADA | Month 12
  Immunogenicity profile of sc remsima®, consisting on the percentage of positive ADA at 12 months
Infliximab trough levels | Month 6
  Immunogenicity profile of sc remsima®, consisting on the course of infliximab trough levels between the inclusion visit and the 6 months visit
Infliximab trough levels | Month 12
  Immunogenicity profile of sc remsima®, consisting on the course of infliximab trough levels between the inclusion visit and the 12 months visit.
Presence or absence of inflammatory flare since the last infusion | Month 3
  Parameter measuring disease activity between the inclusion visit and the 3 months visit
Presence or absence of inflammatory flare since the last infusion | Month 6
  Parameter measuring disease activity between the inclusion visit and the 6 months visit
Presence or absence of inflammatory flare since the last infusion | Month 12
  Parameter measuring disease activity between the inclusion visit and the 12 months visit
Number of flares of disease | Month 3
  Parameter measuring disease activity between the inclusion visit and the 3 months visit
Number of flares of disease | Month 6
  Parameter measuring disease activity between the inclusion visit and the 6 months visit
Number of flares of disease | Month 12
  Parameter measuring disease activity between the inclusion visit and the 12 months visit
Scale of global appreciation of the activity (by the patient) | Month 3
  Scale of global appreciation of the activity (patient) : 0 to 100 (0 = lowest activity, 100 = highest activity) Parameter measuring disease activity between the inclusion visit and the 3 months visit
Scale of global appreciation of the activity (by the patient) | Month 6
  Scale of global appreciation of the activity (patient) : 0 to 100 (0 = lowest activity, 100 = highest activity) Parameter measuring disease activity between the inclusion visit and the 6 months visit
Scale of global appreciation of the activity (by the patient) | Month 12
  Scale of global appreciation of the activity (patient) : 0 to 100 (0 = lowest activity, 100 = highest activity) Parameter measuring disease activity between the inclusion visit and the 12 months visit
Scale of global appreciation of the activity (by the investigator) | Month 3
  Scale of global appreciation of the activity (by the investigator) : 0 to 100 (0 = lowest activity, 100 = highest activity) Parameter measuring disease activity between the inclusion visit and the 3 months visit
Scale of global appreciation of the activity (by the investigator) | Month 6
  Scale of global appreciation of the activity (by the investigator) : 0 to 100 (0 = lowest activity, 100 = highest activity) Parameter measuring disease activity between the inclusion visit and the 6 months visit
Scale of global appreciation of the activity (by the investigator) | Month 12
  Scale of global appreciation of the activity (by the investigator) : 0 to 100 (0 = lowest activity, 100 = highest activity) Parameter measuring disease activity between the inclusion visit and the 12 months visit
Number of swollen/painful joints (Rheumatoid arthritis patient) | Month 3
  Parameter measuring disease activity between the inclusion visit and the 3 months visit
Number of swollen/painful joints (Rheumatoid arthritis patient) | Month 6
  Parameter measuring disease activity between the inclusion visit and the 6 months visit
Number of swollen/painful joints (Rheumatoid arthritis patient) | Month 12
  Parameter measuring disease activity between the inclusion visit and the 12 months visit
Disease Activity Score DAS28 VS (Rheumatoid arthritis patient) | Month 3
  Parameter measuring disease activity between the inclusion visit and the 3 months visit (< 2.6 remission, 2.6-3.2 low activity, 3.2-5.1 moderate activity, >5.1 strong activity)
Disease Activity Score DAS28 VS (Rheumatoid arthritis patient) | Month 6
  Parameter measuring disease activity between the inclusion visit and the 6 months visit (< 2.6 remission, 2.6-3.2 low activity, 3.2-5.1 moderate activity, >5.1 strong activity)
Disease Activity Score DAS28 VS (Rheumatoid arthritis patient) | Month 12
  Parameter measuring disease activity between the inclusion visit and the 12 months visit (< 2.6 remission, 2.6-3.2 low activity, 3.2-5.1 moderate activity, >5.1 strong activity)
Disease Activity Score DAS28 CRP (Rheumatoid arthritis patient) | Month 3
  Parameter measuring disease activity between the inclusion visit and the 3 months visit (< 2.6 remission, 2.6-3.2 low activity, 3.2-5.1 moderate activity, >5.1 strong activity)
Disease Activity Score DAS28 CRP (Rheumatoid arthritis patient) | Month 6
  Parameter measuring disease activity between the inclusion visit and the 6 months visit (< 2.6 remission, 2.6-3.2 low activity, 3.2-5.1 moderate activity, >5.1 strong activity)
Disease Activity Score DAS28 CRP (Rheumatoid arthritis patient) | Month 12
  Parameter measuring disease activity between the inclusion visit and the 12 months visit (< 2.6 remission, 2.6-3.2 low activity, 3.2-5.1 moderate activity, >5.1 strong activity)
BASDAI : Bath Ankylosing Spondylitis Disease Activity Index (Ankylosing Spondylitis patient) | Month 3
  Score : 0 to 100 (0 = lowest activity, 100 = highest activity) Parameter measuring disease activity between the inclusion visit and the 3 months visit
BASDAI : Bath Ankylosing Spondylitis Disease Activity Index (Ankylosing Spondylitis patient) | Month 6
  Score : 0 to 100 (0 = lowest activity, 100 = highest activity) Parameter measuring disease activity between the inclusion visit and the 6 months visit
BASDAI : Bath Ankylosing Spondylitis Disease Activity Index (Ankylosing Spondylitis patient) | Month 12
  Score : 0 to 100 (0 = lowest activity, 100 = highest activity) Parameter measuring disease activity between the inclusion visit and the 12 months visit
Ankylosing Spondylitis Disease Activity Score with CRP (ASDAS-CRP) (Ankylosing Spondylitis patient) | Month 3
  Parameter measuring disease activity between the inclusion visit and the 3 months visit (< 1.3 inactive disease, 1.3-2.1 low activity, 2.1-3.5: high activity, > 3.5 very high activity)
Ankylosing Spondylitis Disease Activity Score with CRP (ASDAS-CRP) (Ankylosing Spondylitis patient) | Month 6
  Parameter measuring disease activity between the inclusion visit and the 6 months visit (< 1.3 inactive disease, 1.3-2.1 low activity, 2.1-3.5: high activity, > 3.5 very high activity)
Ankylosing Spondylitis Disease Activity Score with CRP (ASDAS-CRP) (Ankylosing Spondylitis patient) | Month 12
  Parameter measuring disease activity between the inclusion visit and the 12 months visit (< 1.3 inactive disease, 1.3-2.1 low activity, 2.1-3.5: high activity, > 3.5 very high activity)

CONTACTS AND LOCATIONS:
Overall Officials: Yannick ALLANORE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Rheumatology Department, Cochin Hospital, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: No